CLINICAL TRIAL: NCT01299753
Title: Clinical and Molecular Effects of Catecholamine Blockade Post-burn
Brief Title: Catecholamine Blockade Post-burn
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Marc Jeschke, Principal Investigator, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Propran_Jeschke
Record Dates: First submitted 2011-01-24; First posted 2011-02-18 (Estimated); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Burns
MeSH Terms: conditions — Burns | interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator)
  Interventions: Drug: placebo
- Beta blockade (Experimental)
  Interventions: Drug: propranolol

INTERVENTIONS:
Drug: placebo — identically packed placebo
  Arms: Control
Drug: propranolol — 20-40 mg q6-8h
  Arms: Beta blockade

SUMMARY:
Severe burn is associated with a wide array of stress, metabolic, and physiologic processes in an attempt to restore homeostasis. The catecholamine induced stress response following severe burns is particularly exaggerated and manifests detrimentally as inflammation, insulin resistance, hypermetabolism, and associated profound protein catabolism. The investigators hypothesize that catecholamine blockade will lead to restored IR signaling and result in improved post-burn morbidity. The investigators will further determine the molecular mechanisms mediating these effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 90 years of age
* >25% TBSA burn

Exclusion Criteria:

* Death upon admission
* Decision not to treat due to burn injury severity

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-02; Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Perform oral glucose tolerance test | Conduct at week 1 post admission
  Standard fasting oral glucose tolerance test with an intake of 75 g of glucose. Subsequent measurements (in mg/dl) of glucose in blood, insulin and c-peptide will be conducted over 2 hours.
Perform oral glucose tolerance test | Conduct at week 3 post admission
  Standard fasting oral glucose tolerance test with an intake of 75 g of glucose. Subsequent measurements (in mg/dl) of glucose in blood, insulin and c-peptide will be conducted over 2 hours.
Perform oral glucose tolerance test | Conduct at discharge (1-4 months post admission depending on severity of injury)
  Standard fasting oral glucose tolerance test with an intake of 75 g of glucose. Subsequent measurements (in mg/dl) of glucose in blood, insulin and c-peptide will be conducted over 2 hours.

SECONDARY OUTCOMES:
Measure concentrations of serum cytokines | weekly until discharge (1-4 months post admission depending on severity)
  Inflammatory response will be assessed by measuring the concentrations (pg/ml) of a panel of serum cytokines (IL-1, IFN, TNF etc.) using the Bio-Plex 17-Plex Suspension assay.
Record the episodes of Pneumonia | daily until discharge (1-4 months post admission depending on severity)
  Pneumonia is defined by the following criteria: new progressive and persistent infiltrate, consolidation, or cavitations, in light of the baseline evaluation for inhalational injury on chest X-ray, along with signs of sepsis, worsening gas exchange (decreased P/F ratio), increased O2, and change in the sputum, e.g. purulent or increased sputum production.
Record the episodes of sepsis | daily until discharge (1-4 months post admission depending on severity of injury)
  Patients are evaluated daily and the number of episodes of sepsis or bloodstream infection will be recorded
Measure the levels of activated signaling proteins using protein blotting | assess at 1st operation (week 1-2 post admission on average) and 3rd operation (week 3-4 post admission on average)
  The level of activation of a protein signaling cascade (fold change compared to control), as indicated by the amount of phosphorylated protein substrates (e.g. p-Akt/Akt), will be measured in tissue obtained at operation using protein blotting techniques in the laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: Marc G Jeschke, MD PhD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Ross Tilley Burn Centre - Sunnybrook HSC, Toronto, Ontario, Canada